CLINICAL TRIAL: NCT06316817
Title: Prediction of Hypotension After Induction of General Anesthesia Using Wearable Carotid Artery Doppler Ultrasound Patch in Adult Patients Undergoing Elective Noncardiac Surgery: a Prospective Observational Study
Brief Title: FloPatch for Prevention of Hypotension After Induction of General Anesthesia
Acronym: HI-CAP
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0184-E
Record Dates: First submitted 2024-02-27; First posted 2024-03-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Hypotension on Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FloPatch — A novel, hands-free ultrasound patch for continuous monitoring of quantitative Doppler in the carotid artery.

SUMMARY:
This study is being conducted to find out if a special device called FloPatch™, which sticks to a persons skin and uses ultrasound to check the blood flow in their neck, can tell if someone going to have low blood pressure after they get put to sleep for surgery. The investigators will be testing this in adults who are having elective non-heart surgery. Basically, the goal is to see if this device can help predict who might have low blood pressure during surgery.

Hypotension is a common side-effect of general anesthesia induction, and is related to adverse outcomes, including significantly increasing risk of one-year mortality. Even short durations of intraoperative hypotension have been associated with acute kidney injury (AKI) and myocardial injury. Myocardial injury after non-cardiac surgery (MINS) is a common postoperative complication associated with adverse cardiovascular outcomes, and intraoperative hypotension is believed to be involved in its development.

In the preoperative setting, a systematic review of 50 studies (2,260 patients) evaluating techniques to assess adult patients with refractory hypotension or signs of organ hypoperfusion found that half of all patients were fluid-responsive, pointing to volume status as a significant risk factor, while also presenting a challenge in distinguishing fluid-responders from non-responders. For surgical patients, preoperative fasting, hypertonic bowel preparations, anesthetic agents, and positive pressure ventilation all contribute to reduced effective circulating blood volume. Optimized fluid therapy remains the cornerstone of treatment of hypovolemia, with excellent effectiveness. Since the liberal use of fluids may result in fluid overload, which is associated with the development of pulmonary edema, wound infection, postoperative ileus, and anastomotic leakage, it is imperative to identify those patients who may benefit from it.

The hypothesis is that the corrected Flow Time (cFT) measured by the FloPatch will help predict hypotension after the induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* Undergoing elective noncardiac under general anesthesia

Exclusion Criteria:

* Hypotension, defined as Mean Arterial Pressure (MAP) below 65 mmHg preoperatively on the day of surgery.
* Treated with angiotensin converting enzyme inhibitors (ACE-I) or angiotensin receptor blockers (ARB) on the day of surgery.
* Patients with heart failure with ejection fraction (EF) < 40%.
* A history of any previous neck surgery or trauma.
* Cardiac rhythm other than sinus at the time of common carotid artery corrected Flow Time (cFT) assessment.
* Patients who will receive neuraxial blockade (epidural or spinal) performed before induction of general anesthesia.
* Planned placement of a jugular central venous catheter or surgery to be performed in the area of the FloPatch.
* Patient is pregnant or is undergoing obstetrical surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are adult patients undergoing elective noncardiac surgery at Mount Sinai Hospital in Toronto, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Prognostic ability of preoperative common carotid artery corrected Flow Time (cFT) measurement to predict Post Induction Hypotension(PIH). | within 20 minutes after induction
  The primary outcome is the performance characteristics of the preoperative common carotid artery corrected Flow Time (cFT) to predict Post Induction Hypotension(PIH). PIH will be defined as MAP below an absolute threshold of 65 mmHg or relative threshold of 25% decrease from baseline4 (defined as the first preoperative blood pressure measurement on the morning of surgery), within 20 minutes after induction.

SECONDARY OUTCOMES:
Passive leg raising (PLR) in predicting Post Induction Hypotension(PIH). | The duration of the surgery
  To determine the ability of the change in common carotid artery corrected Flow Time(cFT) during passive leg raising (PLR) and after PLR in predicting Post Induction Hypotension(PIH).
Thresholds of common carotid artery corrected Flow Time (cFT) change during Passive Leg Raising (PLR) in predicting Post Induction Hypotension (PIH). | The duration of the surgery.
  To determine the optimal thresholds for a preoperative common carotid artery corrected Flow Time (cFT) change during PLR, in predicting Post Induction Hypotension(PIH).
Thresholds of common carotid artery corrected Flow Time (cFT) change after Passive Leg Raising(PLR) in predicting Post Induction Hypotension (PIH). | The duration of the surgery.
  To determine the optimal thresholds for a preoperative common carotid artery corrected Flow Time(cFT), after Passive Leg Raising (PLR) in predicting Post Induction Hypotension (PIH).
Time required to get common carotid artery corrected Flow Time(cFT) data. | The duration of the surgery.
  To assess the time required to acquire preoperative common carotid artery corrected Flow Time(cFT) data in patients presenting to surgery.
Common carotid artery corrected Flow Time (cFT) during induction correlation with Post Induction Hypotension(PIH). | The duration of the surgery.
  To determine if common carotid artery corrected Flow Time(cFT) measurements taken during the time of anesthetic induction correlate with the occurrence of Post Induction Hypotension(PIH).

CONTACTS AND LOCATIONS:
Overall Officials: James Khan, MD, Principal Investigator — Staff Anesthesiologist
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No